CLINICAL TRIAL: NCT05272605
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Dose-escalation Study of Adjuvanted SARS-CoV-2 (COVID-19) Beta Variant RBD Recombinant Protein (DoCo-Pro-RBD-1 + MF59®) and mRNA (MIPSCo-mRNA-RBD-1) Vaccines in Healthy Adults Aged 18 to 64 Years Previously Vaccinated With 3 Doses of Licensed SARS-CoV-2 Ancestral Strain Vaccines
Brief Title: Safety and Immune Response of Adjuvanted SARS-CoV-2 (COVID-19) Beta Variant RBD Recombinant Protein (DoCo-Pro-RBD-1 + MF59®) and mRNA (MIPSCo-mRNA-RBD-1) Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Southern Star Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UoM-SARS-CoV-2-01
Record Dates: First submitted 2022-03-03; First posted 2022-03-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — MF59 oil emulsion; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1) 5mcg + MF59 (Experimental): DoCo-Pro-RBD-1 antigen 5mcg mixed with MF59 adjuvant in 0.5 mL suspension, administered intramuscularly in a one dose regimen, on Day 1
  Interventions: Biological: Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1 + MF59)
- Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1)15mcg + MF59 (Experimental): DoCo-Pro-RBD-1 antigen 15mcg mixed with MF59 adjuvant in 0.5 mL suspension, administered intramuscularly in a one dose regimen, on Day 1
  Interventions: Biological: Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1 + MF59)
- Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1) 45mcg + MF59 (Experimental): DoCo-Pro-RBD-1 antigen 45mcg mixed with MF59 adjuvant in 0.5 mL suspension, administered intramuscularly in a one dose regimen, on Day 1
  Interventions: Biological: Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1 + MF59)
- SARS-CoV-2 beta variant RBD mRNA vaccine (MIPSCo-mRNA-RBD-1) 10mcg (Experimental): MIPSCo-mRNA-RBD-1 antigen 10mcg administered intramuscularly as a 0.5 mL dose in a one dose regimen on Day 1
  Interventions: Biological: SARS-CoV-2 beta variant RBD mRNA vaccine
- SARS-CoV-2 beta variant RBD mRNA vaccine (MIPSCo-mRNA-RBD-1) 20mcg (Experimental): MIPSCo-mRNA-RBD-1 antigen 20mcg administered intramuscularly as a 0.5 mL dose in a one dose regimen on Day 1
  Interventions: Biological: SARS-CoV-2 beta variant RBD mRNA vaccine
- SARS-CoV-2 beta variant RBD mRNA vaccine (MIPSCo-mRNA-RBD-1) 50mcg (Experimental): MIPSCo-mRNA-RBD-1 antigen 50mcg administered intramuscularly as a 0.5 mL dose in a one dose regimen on Day 1
  Interventions: Biological: SARS-CoV-2 beta variant RBD mRNA vaccine
- Normal saline (0.9%) (Placebo Comparator): Normal saline (0.9%) administered intramuscularly as a 0.5 mL dose in a one dose regimen on Day 1
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1 + MF59) — Single booster dose in healthy adults previously vaccinated with two doses of CominartyTM (BNT162b2 [mRNA]) or VaxzevriaTM (ChAdOx1-S) COVID-19 and a third booster dose of either ComirnatyTM or SpikevaxTM vaccines.
  Arms: Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1) 45mcg + MF59; Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1) 5mcg + MF59; Adjuvanted SARS-CoV-2 beta variant RBD recombinant protein vaccine (DoCo-Pro-RBD-1)15mcg + MF59
Biological: SARS-CoV-2 beta variant RBD mRNA vaccine — Single booster dose in healthy adults previously vaccinated with two doses of CominartyTM (BNT162b2 [mRNA]) or VaxzevriaTM (ChAdOx1-S) COVID-19 and a third booster dose of either ComirnatyTM or SpikevaxTM vaccines.
  Arms: SARS-CoV-2 beta variant RBD mRNA vaccine (MIPSCo-mRNA-RBD-1) 10mcg; SARS-CoV-2 beta variant RBD mRNA vaccine (MIPSCo-mRNA-RBD-1) 20mcg; SARS-CoV-2 beta variant RBD mRNA vaccine (MIPSCo-mRNA-RBD-1) 50mcg
Other: Normal Saline — Placebo comparator
  Arms: Normal saline (0.9%)

SUMMARY:
This is a study of two experimental SARS-CoV-2 vaccines against the virus called SARS-CoV-2 virus. The first of the experimental vaccines is called DoCo-Pro-RBD-1 + M59® and contains a laboratory made protein which looks the same as a protein in the SARS-CoV-2 virus. As this protein is so similar to a protein in the SARS-CoV-2 virus, it allows the immune system to develop immunity against the real virus by producing specific antibodies against this protein. Antibodies are substances in the blood which could help protect against future infection. The second of the experimental vaccines that will be tested is called MIPSCo-mRNA-RBD-1. This type of vaccine uses messenger ribonucleic acid (mRNA) which is a set of instructions for a cell to make a viral protein called an antigen. Antigens are substances that can trigger the body's defences to produce antibodies that fight against the disease.

This study will test these two experimental COVID-19 vaccines in people who have previously received two doses of ComirnatyTM (Pfizer Australia Pty Ltd) or VaxzevriaTM (AstraZeneca Pty Ltd) and a third booster vaccination with either ComirnatyTM or SpikevaxTM (Moderna). This study is the first time this recombinant protein vaccine and this mRNA vaccine will be given to humans. The purpose of this study is to determine what amount, or dose, of the experimental vaccines is safe and produces the desired immune response and antibody level for future investigations. It will do this by testing 3 different dose levels for each of the two vaccines. Each participant will receive a single vaccine at one of the three dose levels, or a placebo injection. This study is the first time this recombinant protein vaccine and this mRNA vaccine will be given to humans.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, dose-escalation, first-in-human study to assess the safety, reactogenicity and immunogenicity of SARS-CoV-2 beta variant DoCo-Pro-RBD-1 + MF59® and MIPSCo-mRNA-RBD-1 vaccine at three dose levels, administered intramuscularly (IM) as a single booster dose in healthy adults previously vaccinated with two doses of CominartyTM (BNT162b2 [mRNA]) or VaxzevriaTM (ChAdOx1-S) COVID-19 and a third booster dose of either ComirnatyTM or SpikevaxTM vaccines. The study will comprise a Dose-Escalation Phase and an Expanded Phase.

The study vaccines, DoCo-Pro-RBD-1 + MF59®, MIPSCo-mRNA-RBD-1 or placebo (normal saline) will be administered IM in the deltoid region of the upper arm.

The study will enroll healthy adults aged 18 to 64 years of age inclusive. Participants in both the Dose-Escalation Phase and Expanded Phase of the study will be stratified by prior primary course COVID-19 vaccination with CominartyTM or VaxzevriaTM.

ELIGIBILITY:
Inclusion criteria:

To be eligible for this study, participants must meet ALL of the following inclusion criteria:

1. Adults 18 to 64 years of age, inclusive at screening previously vaccinated with a 2-dose schedule of Cominarty™ or Vaxzevria™.
2. ≥ 3 months (90 days) since receipt of a booster dose of either ComirnatyTM or SpikevaxTM.
3. Be in good health as determined by medical history, physical examination, vital signs, and clinical laboratory assessments with no clinically significant abnormalities as judged by the Investigator at screening and randomisation. Vital signs must be within medically acceptable ranges prior to the first vaccination.
4. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea of at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from at least 28 days prior to enrollment and through the end of the study:

   a. Condoms (male or female); Diaphragm; Cervical cap; Intrauterine device; Oral or patch contraceptives; Norplant®, Depo-Provera®, or another regulatory approved contraceptive method; Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle.
5. NOTE: Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post- ovulation methods) and withdrawal method (coitus interruptus) are not acceptable forms of contraception.
6. Agrees to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.
7. Willing and able to give informed consent prior to study enrollment and to comply with all study procedures.

Exclusion criteria:

Potential study participants will be excluded from the study if ANY of the following criteria apply:

1. History of test-confirmed (by PCR, rapid antigen test (RAT) to SARS-CoV-2) COVID-19 infection within 3 months (90 days) prior to randomisation.
2. Participants with a BMI > 35kg/m2.
3. Positive result for rheumatoid factor (RF) at Screening.
4. Positive test at Screening for human immunodeficiency virus (Types 1 or 2) antibody, hepatitis B surface antigen or hepatitis C virus antibody.
5. Clinical laboratory test results not within normal range and judged to be clinically relevant abnormalities by the investigator.
6. History of prior cardiac inflammatory disease (endocarditis, myocarditis or pericarditis).
7. History of demyelinating disease or Guillain Barré syndrome.
8. Fever (non-axillary temperature >37.5°C) or any other symptoms of infection that have not completely resolved within 3 days prior to Randomisation (Day 1).
9. Presence of current active viral infection or bacterial infection, at Screening or Randomisation (Day 1), which is determined by the Investigator to be of clinical significance.
10. Participation in research involving receipt of an investigational product (drug/biologic/device) within 90 days prior to the first study vaccination or an intention to participate in another clinical trial at any time during the conduct of this study.
11. Received any other vaccine within 30 days prior to the first study vaccination, other than licensed influenza vaccine, which can be administered up to 14 days prior to randomization.
12. Any known allergies to products contained in the investigational products.
13. Any history of anaphylaxis to any prior vaccine, food, drug, toxin or other exposure.
14. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.

    NOTE: Stable endocrine disorders (e.g., thyroiditis, pancreatitis), including stable diabetes mellitus with no history of diabetic ketoacidosis) are NOT excluded.
15. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to first study vaccination.

    NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10mg of prednisone per day or equivalent. The use of topical or intranasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted.
16. Received immunoglobulin, blood-derived products, or immunosuppressant drugs or donation of blood/blood products within 90 days prior to vaccination or planned receipt or donation during the study period.
17. Thrombocytopaenia, contraindicating intramuscular vaccination, based on the Investigator's judgment.
18. Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination based on the Investigator's judgement.
19. Active cancer (malignancy) on therapy within one year prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo malignancy and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the Investigator).
20. Participants who are breastfeeding, pregnant or who plan to become pregnant prior to the end of study.
21. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the first study vaccine dose that, in the opinion of the Investigator, might interfere with protocol compliance.
22. Have a tattoo/scar/birthmark or any other skin condition affecting the deltoid area that may, in the Investigator's opinion, interfere with injection site assessments.
23. Any other condition that, in the opinion of the Investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the trial vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
24. Study team member or immediate family member of any study team member (inclusive of Sponsor, Contract Research Organization (CRO), and study site personnel involved in the conduct or planning of the study).
25. Aboriginal and Torres Strait Islander person aged 50 years or older.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Serious adverse events (SAEs), medically attended adverse events (MAAEs) and any adverse events (AEs) leading to study withdrawal at any time during the study. | Through to study completion at Day 181.
  Frequency
SAEs post vaccination. | Day 1 to 29 (28 Days post vaccination).
  Frequency
Solicited local and systemic reactogenicity AEs post vaccination. | Within 7 days after vaccination (Day 1)
  Frequency, severity, duration and peak intensity
Unsolicited AEs post vaccination. | Day 1 to Day 29 (28 days post vaccination).
  Frequency
Percentage of participants who achieve a boost response post vaccination. | 28 days after vaccination
  Defined as a 4-fold increase in SARS-CoV-2 neutralising or RBD-specific Ab titres from baseline.

SECONDARY OUTCOMES:
MAAEs from Day 1 to 6 months after vaccination. | 6 months after vaccination.
  MeDRA classification, severity score and relatedness.
The number of participants that develop an antibody response at least 4 times higher than baseline antibody titers. | At baseline (Day 1), Day 29 (28 days after vaccination), and 3, and 6 months after vaccination
  Number of participants that develop an antibody response at least 4 times higher than baseline antibody titers (before injection of the vaccine candidate or placebo), as assessed using in vitro ELISA assays for binding of the SARS-CoV-2 RBD to ACE2, and neutralising antibody assays that measure the ability to block RBD binding to ACE-2 or the ability of virus to infect cells in vitro). The magnitude and durability of those antibody responses over time will also be used to indicate the strength of the response within each participant to each vaccine in each cohort, and in relation to which vaccine the participants had previously received, compared to those participants that received placebo.
Number of participants that mount a T cell response for SARS-CoV-2 RBD-derived peptide antigens. | Baseline (Day 1), Day 8 (7 days after vaccination), Day 29 (28 days after vaccination) and 3 and 6 months after vaccination.
  Number of participants that develop a T cell response in the short term (Day 8) and in the longer term (Day 29, 3 and 6 months after vaccination) in response to the vaccine candidate compared to their baseline (Day 1) T cell responses. T cell responses will be measured by flow cytometry looking for activated CD4 and CD8 T cells, including the percentage of T cells that respond to peptide antigens derived from the SARS-CoV-2 RBD. The magnitude and durability of those T cell responses over time will also be used to indicate the strength of the response within each participant to each vaccine in each cohort, and in relation to which vaccine the participants had previously received, compared to those participants that received placebo.
Number of participants that mount a T cell response that leads to type-1 cytokines (such as Interferon-gamma) versus type-2 cytokines (such as Interleukin 4, 5 and 13). | Baseline (Day 1), Day 8 (7 days after vaccination), Day 29 (28 days after vaccination) and 3 and 6 months after vaccination.
  For participants that develop a T cell response, two types of T cell response will be assessed, based on whether the activated T cells produce the cytokine Interferon-gamma, indicative of a type 1 cytokine response, or Interleukins 4, 5 and 13, indicative of a type 2 cytokine response. Cytokines will be measured following T cell activation with SARS-CoV-2-derived peptide antigens in vitro, using assays for cytokines will include intracellular cytokine staining as measured by flow cytometry, and elispot, as measured by an elispot reader.
The ratio of T cell derived type 1 versus type 2 cytokines in participants that mount a T cell response. | Baseline (Day 1), Day 8 (7 days after vaccination), Day 29 (28 days after vaccination) and 3 and 6 months after vaccination.
  For participants that develop a T cell response, the ratio of type 1 cytokine to type 2 cytokines, measured by intracellular cytokine staining and by ELISpot, will be determined for at each timepoint, compared to placebo controls and baseline responses.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Terry Nolan, Principal Investigator — Peter Doherty Institute for Infection and Immunity, The University of Melbourne
Locations (2):
- Australia (2):
  - Vaccine and Immunisation Research Group, Doherty Institute, University of Melbourne, Melbourne, Victoria
  - Royal Melbourne Hospital, Victorian Infectious Diseases Service (VIDS), Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nolan TM, Deliyannis G, Griffith M, Braat S, Allen LF, Audsley J, Chung AW, Ciula M, Gherardin NA, Giles ML, Gordon TP, Grimley SL, Horng L, Jackson DC, Juno JA, Kedzierska K, Kent SJ, Lewin SR, Littlejohn M, McQuilten HA, Mordant FL, Nguyen THO, Soo VP, Price B, Purcell DFJ, Ramanathan P, Redmond SJ, Rockman S, Ruan Z, Sasadeusz J, Simpson JA, Subbarao K, Fabb SA, Payne TJ, Takanashi A, Tan CW, Torresi J, Wang JJ, Wang LF, Al-Wassiti H, Wong CY, Zaloumis S, Pouton CW, Godfrey DI. Interim results from a phase I randomized, placebo-controlled trial of novel SARS-CoV-2 beta variant receptor-binding domain recombinant protein and mRNA vaccines as a 4th dose booster. EBioMedicine. 2023 Dec;98:104878. doi: 10.1016/j.ebiom.2023.104878. Epub 2023 Nov 27. PMID 38016322
- See also: Broad immunity to SARS-CoV-2 variants of concern mediated by a SARS-CoV-2 receptor-binding domain protein vaccine — https://www.medrxiv.org/content/10.1101/2022.08.05.22278425v1